CLINICAL TRIAL: NCT01661712
Title: Randomised, Double-blinded, Sham-controlled Cross-over Trial of Continuous Transcutaneous Electrical Stimulation of the Pharyngeal Dilator Muscles in Obstructive Sleep Apnoea
Brief Title: Continuous Transcutaneous Electrical Stimulation in Sleep Apnoea
Acronym: TESLA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Joerg Steier, MD, PhD, Guy's and St Thomas' NHS Foundation Trust
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SOSATS2012-V1.0-01/08/2012
Record Dates: First submitted 2012-08-02; First posted 2012-08-09 (Estimated); Results first posted 2018-11-02 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-11

CONDITIONS: Obstructive Sleep Apnoea
Keywords: obstructive sleep apnoea,; continuous transcutaneous electrical stimulation
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transcutaneous electrical stimulation (Active Comparator): One night of transcutaneous electrical stimulation (electrical current titrated according to skin sensation)
  Interventions: Device: Transcutaneous electrical stimulation
- Sham stimulation (Sham Comparator): One night of sham stimulation (no electrical current)
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Transcutaneous electrical stimulation — Transcutaneous electrical stimulation (one night of electrical current titrated according to skin sensation)
  Arms: Transcutaneous electrical stimulation
Device: Sham stimulation — Sham stimulation for one night (no electrical stimulation)
  Arms: Sham stimulation

SUMMARY:
The aim of this randomized, double-blinded, sham-controlled cross-over trial is to demonstrate the effectiveness of continuous transcutaneous electrical stimulation of the pharyngeal dilator muscles to reduce sleep-disordered breathing.

DETAILED DESCRIPTION:
Obstructive sleep apnoea is the most common problem of sleep-disordered breathing. It affects at least four percent of the male and two percent of the female adult population. It is associated with excessive daytime sleepiness, causing significant disturbance of daytime routines affecting work, social life and memory; untreated, it also causes a significant cardiovascular and metabolic risk. The best available treatment for obstructive sleep apnoea is continuous positive airway pressure (CPAP). However, not everyone eligible tolerates this treatment because it requires them to sleep with a nasal or full-face mask that is connected by a tube to a machine. Although CPAP is recommended by the National Institute for Health and Clinical Excellence (NICE) for moderate-severe sleep apnoea, approximately one third of sleep apnoea patients who should be on CPAP stop therapy within five years. Mild sleep apnoea is currently treated with mandibular advancement splints and generic sleep hygiene advice.

Continuous transcutaneous electrical stimulation (CTES) of the submental region activates the muscles that dilate the upper airway. This is where airway obstruction occurs in sleep apnoea. It has been shown that CTES at night for short periods (10minutes) effectively stimulates the genioglossus muscle, the strongest pharyngeal dilator and reduces upper airway obstruction, work of breathing and neural respiratory drive in patients with sleep apnoea. The London Respiratory Muscle Groups, based within King's Health Partners and the Royal Brompton Hospital, has developed a CTES stimulator device. This device senses apnoeas and snoring and delivers CTES until normal ventilation has been restored.

We propose to undertake a randomized, double-blinded, sham-controlled cross-over trial with sleep apnoea patients to evaluate the efficacy of this method. Patients will be randomly assigned to a night of CTES or sham-stimulation. The primary outcome measure is the number of oxygen desaturations per hour (ODI) caused by apnoeas and the secondary outcome measures are sleepiness, as measured by the Epworth sleepiness score, the apnoea-hypopnoea-index (AHI) and comfort, as assessed by a visual analogue score. The sample size Calculation using data from our own published pilot study revealed that this study would require 44 patients to be enroled. The mean study duration until all outcomes will be assessed for each patient will be four weeks. We plan to commence the study in winter 2012/13 for a period of two years, including analysis and publication, to be concluded in December 2014.

ELIGIBILITY:
Inclusion Criteria:

* males and females, age >18years and <75years, body-mass index (BMI) >18 and <40kg/m2, non-smokers, sleep apnoea with an ODI ≥15/h or sleep apnoea with an ODI ≥5/h plus an Epworth sleepiness score >10.

Exclusion Criteria:

* morbid obesity (BMI>40kg/m2) or cachexia (BMI<18kg/m2), obesity-hypoventilation syndrome (total sleep time with oxygen saturation (SpO2) less than 90% of more than 10% of the night), active smokers or smoking history of >20pack years, acute or critical illness, acute psychosis or chronic mental disorder affecting capacity, previous home-mechanical non-invasive ventilation and metal implants in the upper part of the body (this excludes dental implants).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2013-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joerg Steier, MD, PhD, Principal Investigator — Guy´s & St Thomas´ NHS Foundation Trust
Locations (1):
- Guy´s & St Thomas´ NHS Foundation Trust, London, United Kingdom

REFERENCES:
- [Result] Steier J, Seymour J, Rafferty GF, Jolley CJ, Solomon E, Luo Y, Man WD, Polkey MI, Moxham J. Continuous transcutaneous submental electrical stimulation in obstructive sleep apnea: a feasibility study. Chest. 2011 Oct;140(4):998-1007. doi: 10.1378/chest.10-2614. Epub 2011 Mar 31. PMID 21454399
- [Derived] Pengo MF, Xiao S, Ratneswaran C, Reed K, Shah N, Chen T, Douiri A, Hart N, Luo Y, Rafferty GF, Rossi GP, Williams A, Polkey MI, Moxham J, Steier J. Randomised sham-controlled trial of transcutaneous electrical stimulation in obstructive sleep apnoea. Thorax. 2016 Oct;71(10):923-31. doi: 10.1136/thoraxjnl-2016-208691. Epub 2016 Jul 19. PMID 27435610
- See also: Guy's & St Thomas' National Health Service (NHS) Foundation Trust homepage — http://www.gstt.nhs.uk

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a randomised, sham-controlled crossover trial using transcutaneous electrical stimulation of the upper airway dilator muscles in patients with confirmed obstructive sleep apnea (OSA).
Pre-assignment Details: A total of 390 patients were assessed, 44 patients were screened. 8 patients were excluded as screening failures. 36 patients were randomised into the sequence 'Sham Stimulation, then True Stimulation' (n=18) or 'True Stimulation, then Sham Stimulation' (n-18). All 36 randomised subjects completed the trial, serving as their own control.
Groups:
- Sham Stimulation, Then True Stimulation: The patient will 1st undergo a sleep study with Sham stimulation. An identical setup to the intervention will be used with the software indicating stimulation to keep staff blinded to the intervention.
  Then patients will undergo a washout period (>3nights) and return for a 2nd sleep study on true stimulation to complete the trial.
  Transcutaneous electrical stimulation (SOSATS device, MORGAN Innovation&Technology Ltd., Petersfield, UK):
  The SOSATS unit is a first generation sleep apnoea research device which is programmed and controlled by an external personal computer (PC) or laptop via a visual interface. It stimulates the pharyngeal dilator muscles to reduce sleep apnoea.
- Transcutaneous Electrical Stimulation, Then Sham Stimulation: The patient will undergo the 1st sleep study with continuous transcutaneous electrical stimulation.
  Then patients will undergo a washout period (>3nights) and return for a 2nd sleep study on sham stimulation to complete the trial.
  Transcutaneous electrical stimulation (SOSATS device, MORGAN Innovation&Technology ltd., Petersfield, UK):
  The SOSATS unit is a first generation sleep apnoea research device which is programmed and controlled by an external PC or laptop via a visual interface. It stimulates the pharyngeal dilator muscles to reduce sleep apnoea.
Period: Overall Study
Arm/Group | Sham Stimulation, Then True Stimulation | Transcutaneous Electrical Stimulation, Then Sham Stimulation
Started (1st night, patients completed intervention/sham arm in randomised assigned order, cross-over design.) | 18 (initial sham stimulation night) | 18 (initial night on transcutaneous electrical stimulation)
Washout Period (Washout period of >3 nights.) | 18 (>Three nights of no stimulation/sham stimulation) | 18 (>Three nights of no stimulation/sham stimulation)
Completed (2nd night, patients completed intervention/sham arm in randomised assigned order, cross-over design.) | 18 (night on transcutaneous electrical stimulation) | 18 (sham stimulation night)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sham Stimulation First, Then Transcutaneous Electrical Stimula: The patient will undergo a sleep study and continuous transcutaneous electrical stimulation will be administered during the night. After 3 days of wash out the patient will undergo a sleep study with the sham intervention and no continuous transcutaneous electrical stimulation will be administered.
  An identical setup to the intervention will be used with the software indicating stimulation to keep staff blinded to the intervention.
  Transcutaneous electrical stimulation (SOSATS device, MORGAN Innovation&Technology ltd., Petersfield, UK): The SOSATS unit is a first generation sleep apnoea research device which is programmed and controlled by an external PC or laptop via a visual interface.
  It stimulates the pharyngeal dilator muscles in order to reduce sleep apnoea.
- Transcutaneous Electrical Stimulation First, Then Sham Stimula: The patient will undergo a sleep study with Sham stimulation. After 3 days of wash out the patient will will undergo a sleep study and continuous transcutaneous electrical stimulation will be administered during the night An identical setup to the intervention will be used with the software indicating stimulation to keep staff blinded to the intervention.
  Transcutaneous electrical stimulation (SOSATS device, MORGAN Innovation&Technology ltd., Petersfield, UK): The SOSATS unit is a first generation sleep apnoea research device which is programmed and controlled by an external PC or laptop via a visual interface.
  It stimulates the pharyngeal dilator muscles in order to reduce sleep apnoea.
- Total: Total of all reporting groups
Arm/Group | Sham Stimulation First, Then Transcutaneous Electrical Stimula | Transcutaneous Electrical Stimulation First, Then Sham Stimula | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.2 (11.9) | 50.6 (11) | 50.8 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6
  Male | 13 | 17 | 30

OUTCOME MEASURES:

1. Primary Outcome: 4% Oxygen Desaturation Index (ODI, 4%)
Description: The primary outcome measure for this trial is the 4% oxygen desaturation index (ODI, 4%) per hour of sleep (h-1). The 4% ODI was chosen as primary outcome parameter over the AHI because an incomplete re-opening of the upper airway during an ongoing apnoeic effort caused by transcutaneous electrical stimulation (CTES) may result in a nominal increase of the AHI. We consider that the 4% ODI would be a more robust marker for the severity of sleep apnoea, low average oxygen levels indicating obesity-hypoventilation syndrome which will be an exclusion criterion.
  Although a specific cut off is not well defined a 4% ODI ≥5 represent mild OSA whilst a 4% ODI ≥15 represents moderate-severe OSA. Normal range is usually considered 0-5 events/hour.
Time Frame: 1st sleep study compared to 2nd sleep study (randomised order of intervention/sham or sham/intervention)
Measure: Median (Inter-Quartile Range); unit: oxygen desaturation events/hour
Groups:
- Sham Stimulation: patients that underwent the Sham stimulation night study
- Active Treatment: Patients that underwent the stimulation overnight sleep study
Arm/Group | Sham Stimulation | Active Treatment
Number analyzed (Participants) | 36 | 36
oxygen desaturation events/hour | 26.9 [17.5 to 39.5] | 19.5 [11.6 to 40.0]

2. Secondary Outcome: Apnoea-Hypopnoea Index (AHI)
Description: The Apnoea-Hypopnoea Index (AHI) is an index used to indicate the severity of sleep apnea. It is represented by the number of apnea and hypopnea events per hour of sleep. An apnea (pause in breathing) is defined by a temporary cessation of breathing that must last for at least 10 seconds and be associated with a decrease in blood oxygenation. A hypopnoea is a reduction of ventilation (shallow breathing) but not a complete cessation of breathing, lasting al least 10 seconds and associated with a decrease in blood oxygenation.
Time Frame: 1st sleep study compared to 2nd sleep study (randomised order of intervention/sham or sham/intervention)
Measure: Median (Inter-Quartile Range); unit: events/hour
Groups:
- Sham Stimulation: sham stimulation night
- Transcutaneous Electrical Stimulation: Transcutaneous electrical stimulation night
Arm/Group | Sham Stimulation | Transcutaneous Electrical Stimulation
Number analyzed (Participants) | 36 | 36
events/hour | 33.8 [16.6 to 46.1] | 23.7 [11.4 to 47.6]

3. Secondary Outcome: Nadir Oxygenation
Description: The nadir oxygenation (lowest SpO2, %) during the sleep study is measured while the patients are asleep.
Time Frame: 1st sleep study compared to 2nd sleep study (randomised order of intervention/sham or sham/intervention)
Measure: Median (Inter-Quartile Range); unit: % of haemoglobin that is oxygenated
Groups:
- Transcutaneous Electrical Stimulation: Transcutaneous electrical stimulation: the patient will undergo a sleep study and continuous transcutaneous electrical stimulation during the night ("active treatment").
  Transcutaneous electrical stimulation (SOSATS device, MORGAN Innovation&Technology ltd., Petersfield, UK): The SOSATS unit is a first generation sleep apnoea research device which is programmed and controlled by an external PC or laptop via a visual interface.
  It stimulates the pharyngeal dilator muscles in order to reduce sleep apnoea.
- Sham Stimulation: Sham stimulation: the patient will undergo a sleep study with Sham stimulation. An identical setup to the intervention will be used with the software indicating stimulation to keep staff blinded to the intervention (Modes are labelled "A" and "B" for real and sham stimulation and observers will not be able to tell the difference on the screen).
  Sham stimulation (SOSATS device, MORGAN Innovation&Technology ltd., Petersfield, UK): The patient will undergo a sleep study with sham transcutaneous electrical stimulation. The setup will be identical to the intervention, but a blinded mode in the software application will stop triggering electrical current despite indicating on the monitor that stimulation is being applied.
Arm/Group | Transcutaneous Electrical Stimulation | Sham Stimulation
Number analyzed (Participants) | 36 | 36
% of haemoglobin that is oxygenated | 81.0 [74.0 to 84.0] | 80.5 [74.5 to 86.0]

4. Secondary Outcome: Patient Comfort
Description: Patient comfort during the sleep study, as measured by a visual analogue scale (0-10 points). Higher values in the scale range represent a better outcome.
Time Frame: 1st sleep study compared to 2nd sleep study (randomised order of intervention/sham or sham/intervention)
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Transcutaneous Electrical Stimulation | Sham Stimulation
Number analyzed (Participants) | 36 | 36
units on a scale | 6.4 [2.4 to 8.0] | 5.6 [2.9 to 7.1]

5. Secondary Outcome: Device Acceptance
Description: Device acceptance during sleep study, as measured by a visual analogue scale (0-10points). Higher values in the scale range represent a better outcome.
Time Frame: 1st sleep study compared to 2nd sleep study (randomised order of intervention/sham or sham/intervention)
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Sham Stimulation | Active Treatment
Number analyzed (Participants) | 36 | 36
units on a scale | 9.9 [9.5 to 10.0] | 9.9 [9.7 to 10.0]

6. Secondary Outcome: Sleepiness
Description: Daytime sleepiness as an ad-hoc measurement, as measured by the Stanford Sleepiness Scale (0-7 points, x). Higher values in the scale range represent more severe sleepiness.
Time Frame: 1st sleep study compared to 2nd sleep study (randomised order of intervention/sham or sham/intervention)
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Transcutaneous Electrical Stimulation | Sham Stimulation
Number analyzed (Participants) | 36 | 36
units on a scale | 3.0 [2.0 to 3.0] | 3.0 [2.0 to 3.5]

ADVERSE EVENTS:
Arm/Group | Sham Stimulation | Active Treatment
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 1/36 | 1/36
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham Stimulation (N=36) | Active Treatment (N=36)
claustrophobia (Psychiatric disorders) | 1 (1) | 1 (1) — The only significant side effect observed was one patient who complained about claustrophobia at night; this was during both treatment nights

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No